CLINICAL TRIAL: NCT03894605
Title: Assessment ofDermatological Abnrmalities in Beta-thalassemia Major in Assiut University Pediatric Hospital
Brief Title: Dermatological Abnormalities in Beta-thalassemia Major
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Neveen Mamdoh Farag, Principal investigator, Assiut University
Other Study IDs: DBTM
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: thalassemia — thalassemic patient use chelator and thaladssemic patient with frequent blood transfusion

SUMMARY:
to study the frequency and pattern of dermatological abnormalities in egyptian childern with beta thalassemia.relationof abnormalities to duration of disease and frequency of transfusion

DETAILED DESCRIPTION:
thalassemia refers to agroup of inherited disease characterized by decreased or absent synthesis of normal globin .skinvdisorders are usually neglected and frequently underdiagnosed among these patients.skin disease specially pruritus and xerosis are observed highly frequently in patients with beta-thalassemia.pityriasis alba is arelatively common skin disorder.the trophic skin changes and leg ulcers occurred after the age of 15 years

ELIGIBILITY:
Inclusio2n Criteria:

* clinical diagnosis of dermatological abnormalities in thalassemic patient. must be on chelator

Exclusion Criteria:

* patient with other hemolytic anemia. childern with any abnormalities prior to the diagnosis of thalassemi

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: all patient examined by single dermatologist to record any dermatological abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-03-02 (Estimated); Study Completion 2021-04-02 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with dermatological disorders due to iron overload Iron overload cause dermatological abnormalities | one month
  the number of patients who develop any dermatological disorder as a result of iron overload after frequent blood transfusion

REFERENCES:
- [Background] Cao A, Galanello R. Beta-thalassemia. Genet Med. 2010 Feb;12(2):61-76. doi: 10.1097/GIM.0b013e3181cd68ed. PMID 20098328
- [Result] El-Dash H, Adel S. Cutaneous manifestations in Egyptian children with beta-thalassemia major: Relationship with serum ferritin, thyroid profile, and treatment modalities. Pediatr Dermatol. 2018 Sep;35(5):639-643. doi: 10.1111/pde.13570. Epub 2018 Jun 26. PMID 29943859
- [Result] Dogramaci AC, Savas N, Ozer B, Duran N. Skin diseases in patients with beta-thalassemia major. Int J Dermatol. 2009 Oct;48(10):1057-61. doi: 10.1111/j.1365-4632.2009.04176.x. PMID 19785086
- [Result] CHANG PY, KUO CL, KHOO FY. The anatomic distribution of the lesions in pulmonary tuberculosis. Med Abstr. 1945 Oct;63A:237-43. No abstract available. PMID 20997138